CLINICAL TRIAL: NCT03541044
Title: A Single Dose Bioequivalence Study of a 2 mg Prototype Mini Nicotine Lozenge vs 2 mg Nicotine Mini Lozenge (Nicorette Minis) Healthy Smokers Under Fasting Conditions
Brief Title: A Bioequivalence Study of Two Nicotine Lozenges in Fasting Conditions in Healthy Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 207791
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): Participants will receive a single Nicotine Prototype Mini lozenge (2mg) by oral/buccal route of administration.
  Interventions: Drug: Nicotine Prototype Mini lozenge
- Reference Product (Active Comparator): Participants will receive a single Nicorette Mini lozenge (2 mg) by oral/buccal route of administration.
  Interventions: Drug: Nicorette Mini Lozenge

INTERVENTIONS:
Drug: Nicotine Prototype Mini lozenge — A single dose of a prototype nicotine 2mg lozenge will be placed in participants mouth, occasionally moving it side to side. Allowing it to slowly dissolve and try to minimize swallowing. Participants will be instructed not to chew lozenge. The lozenge should be completely dissolved.
  Arms: Test Product
Drug: Nicorette Mini Lozenge — A single dose of a 2 mg nicotine polacrilex mini lozenge (Nicorette Minis) will be placed in participants mouth, occasionally moving it side to side. Allowing it to slowly dissolve and try to minimize swallowing. Participants will be instructed not to chew lozenge. The lozenge should be completely dissolved.
  Arms: Reference Product

SUMMARY:
This study will assess the bioequivalence of the test product (Nicotine Prototype Mini lozenge 2 milligrams [mg]) to a commercial reference product (nicotine polacrilex mini lozenge 2 mg) in healthy smokers under fasting conditions.

DETAILED DESCRIPTION:
This study will be a single center, randomized, open label, single dose, two-way crossover in healthy smokers that smoke their first cigarette more than 30 minutes of waking. This study will consist of following Visits: Visit 1 (Screening), Visit 2 (Study Period 1), followed by a Washout period and Visit 3 (Study Period 2). Each participant will be treated with a single dose of the two study treatments (test and reference) in a randomized sequence. Participants will be confined in the study facility for approximately 60 hours during each study session (for 36 hours pre-dosing and for 24 hours post dosing) during which pharmacokinetic (PK) blood samples will be obtained. Participants are to abstain from smoking during the confinement periods and be subject to random measurements of expired carbon monoxide (CO) to confirm abstinence. The CO levels must be ≤10 parts per million (ppm) throughout the study session. There will be at least 5-day and not more than 7-day clinical furlough period between treatment periods. For each treatment period, the clinical confinement period with restriction of smoking is at least 36 hours prior to dosing.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Healthy participants which is defined as in general good physical health, as judged by the investigator and no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure, respiratory rate, oral body temperature and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Body Mass Index (BMI) of 19 to 27 Kilogram per meter square (kg/m2), inclusive; and a total body weight >50 kg (110 pounds [lbs]).
* Female participants of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 5 days after the last dose of assigned treatment. Female participants who are not of childbearing potential must meet at least one of the following criteria: a) Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state. b) Have undergone a documented hysterectomy and/or bilateral oophorectomy.
* Participant admits to having smoked commercially available cigarettes daily for the preceding 12 months and to routinely smoking his or her first cigarette more than 30 minutes upon awakening. Brief periods of non-smoking (e.g. due to illness, trying to quit, participation in a study where smoking was prohibited) during that time will be permitted at the discretion of the PI (Principal Investigator).

Exclusion Criteria:

* Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Participants who are GSK employees directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s) within 30 days prior to first dose and during study participation.
* Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the Participant inappropriate for entry into this study.
* Pregnant female Participants.
* Breastfeeding female Participants.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Participant has used any nicotine replacement therapy within 21 days prior to the first study session.
* Participant has used chewing tobacco, tobacco products or electronic cigarettes other than cigarettes within 21 days of Visit 1.
* Use of prescription or non-prescription drugs and dietary supplements within two weeks or 5 half-lives, whichever is longer, prior to the first dose of investigational product until the end of the study. Allowed treatments are: Systemic contraceptives and hormone replacement therapy, as long as female Participant is on stable treatment for at least 3 months and continues treatment throughout the study. Evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation.
* History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* A positive urine drug screen for THC, amphetamine, cocaine, 3,4-methylenedioxy-N-methylamphetamine (MDMA)/ecstasy, methamphetamine, or opiates; and urine alcohol testing during screening or baseline testing.
* Participant is unwilling to abstain from tobacco or nicotine-containing product use during each study session (from start of baseline to the completion of the last PK blood sampling). CO measurement immediately prior to randomization (first treatment session) and dosing (second treatment session) should be ≤ 10 parts per million (ppm) for the Participant to be dosed.
* Participant ingests more than 5 cups of coffee or tea a day (or equivalent xanthine consumption using other products).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer).
* A medical history that, in the opinion of the investigator, might jeopardize the safety of the Participant, e.g., recent myocardial infarction or cerebrovascular accident (i.e., within 12 weeks prior to the first study session), severe cardiac arrhythmia, history of seizures, orthostatic hypotension, cardiovascular disease, stroke, or TIA.
* A medical history, which, in the opinion of the investigator, might impact the validity of the study results, may require treatment, or make the Participant unlikely to finish the study.
* Oral surgery within 4 weeks of dosing, dental work or extractions within 2 weeks of dosing, or presence of any clinically significant (as determined by the principal investigator or designee) oral pathology including lesions, sores or inflammation.
* Diagnosis of long QT syndrome or QTc > 460 msec for males and > 470 msec for females at screening.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance including, but not limited to, any of the following: i)Presence of active oesophagitis, oral or pharyngeal ulceration, inflammation, gastritis, gastric ulcer or peptic ulcer or other diseases; ii) Presence of gum disease, xerostomia, dentures or any dental work that could affect the conduct of the study as determined by the investigator or designee; iii) Renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine or urea or the presence of clinically significant abnormal urinary constituents (e.g. albuminuria). Minor deviations of laboratory values from the normal range are permitted, if judged by the investigator to have no clinical relevance; iv) Ongoing hepatic disease or impaired hepatic function at screening. A candidate will be excluded if more than one of the following lab value deviations are found and are clinical ly relevant: aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT), Alanine Aminotransferase/ serum glutamic-pyruvic transaminase (ALT/SGPT), γ-glutamyl transpeptidase (γGGT), alkaline phosphatase, bilirubin or CK. Minor deviations of laboratory values from the normal range are permitted, if judged by the investigator to have no clinical relevance; v) History or clinical evidence at screening of pancreatic injury or pancreatitis; vi) Evidence of urinary obstruction or difficulty in voiding at screening; vii) History of malignancy or neoplastic disease of any organ system (except for localized basal cell skin carcinoma), treated or untreated, within the past 5 years prior to screening, regardless of whether there is evidence of local recurrence or metastases. viii) Clinically relevant chronic or acute infectious illnesses or febrile infections within 2 weeks prior to start of the study (enrollment). ix) Other clinically significant laboratory findings in the opinion of the Investigator at screening.
* A positive serum Hepatitis B surface antigen, Hepatitis C antibodies, or human immunodeficiency virus (HIV) test result.
* Blood: a) Has donated or experienced significant blood loss (470 mL) within 56 days of Visit b) Hemoglobin value < 12.0 grams per deciliter (g/dL).
* Participants who have previously been enrolled in this study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2019-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in United States. A total of 90 participants were screened, of whom 46 were randomized for treatment and 44 were screen failures.
Pre-assignment Details: Participants received treatment in one of the two sequences; treatment A (Prototype Mini Lozenge: Reference drug) followed by treatment B (Nicorette Mini lozenge: Investigational drug) or vice versa in each of the study period 1 and 2.
Groups:
- Prototype-Washout-Nicorette: Participants randomized to this group received a single dose of Treatment A: 2 milligrams (mg) of Prototype Mini Lozenge administered orally on Day 0 in Treatment Period 1. It was followed by a washout period of at least 5 days to a maximum of 7 days, then participants received Treatment B: 2 mg of Nicorette Mini lozenge administered orally on any one day from Day 5-Day 7 (depending upon washout period) in Treatment Period 2. All these doses were administered after an overnight fast of at least 10 hours in each period. Participants were confined in the study facility for approximately 60 hours during each treatment period (for 36 hours predose and for 24 hours postdose) with abstinence from smoking during which they were subjected to random measurements of expired carbon monoxide (CO) to confirm abstinence (CO levels must have been less than or equal to[<=] 10 parts per million [ppm] throughout the treatment period).
- Nicorette-Washout-Prototype: Participants randomized to this group received a single dose of Treatment B: 2 mg of Nicorette Mini lozenge administered orally on Day 0 in Treatment Period 1. It was followed by a washout period of at least 5 days to a maximum of 7 days, then participants received Treatment A: 2 mg of Prototype Mini Lozenge administered orally on any one day from Day 5-Day 7 (depending upon washout period) in Treatment Period 2. All these doses were administered after an overnight fast of at least 10 hours in each period. Participants were confined in the study facility for approximately 60 hours during each treatment period (for 36 hours predose and for 24 hours postdose) with abstinence from smoking during which they were subjected to random measurements of expired CO to confirm abstinence (CO levels must have been <= 10 ppm throughout the treatment period).
Period: Study Period 1: Up to Day 1
Arm/Group | Prototype-Washout-Nicorette | Nicorette-Washout-Prototype
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0
Period: Washout Period: 5 to 7 Days
Arm/Group | Prototype-Washout-Nicorette | Nicorette-Washout-Prototype
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0
Period: Study Period 2: Up to Day 8
Arm/Group | Prototype-Washout-Nicorette | Nicorette-Washout-Prototype
Started | 23 | 23
Completed | 21 | 23
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all randomized participants who received at least one dose of study medication.
Groups:
- All Treatment Combined: All randomized participants received either a single dose of TreatmentA:2mg of Prototype Mini Lozenge administered orally on Day0 in Treatment Period1 followed by TreatmentB:2mg of Nicorette Mini lozenge administered orally on any one day from Day 5-Day 7(depending upon washout period) in Treatment Period2 or vice versa. Washout period was of at least 5days to maximum of 7days between two treatment periods. All these doses were administered after an overnight fast of at least 10 hours in each period. Participants were confined in the study facility for approximately 60 hours during each treatment period (for 36 hours predose and for 24 hours postdose) with abstinence from smoking during which they were subjected to random measurements of expired CO to confirm abstinence (CO levels must have been <=10 ppm throughout the treatment period).
Arm/Group | All Treatment Combined
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Bioequivalence of Prototype Mini Lozenges With Nicorette Mini Lozenge by Measuring Area Under the Plasma Concentration Versus Time Curve From Time Zero to Time t (AUC [0-t])
Description: Bioequivalence of prototype mini lozenges with nicorette mini lozenge was assessed by measuring AUC(0-t), where t= time of the last measurable plasma concentration. AUC(0-t) was calculated using the linear trapezoidal with linear interpolation method. A linear mixed-effects model was fit to the natural log (ln)-transformed PK variable (AUC0-t), as the dependent variable, and treatment, period, and sequence as fixed effects. Participant nested within sequence was a random effect. The treatment difference and its 90% CI were exponentiated to obtain the geometric mean ratios (GMR) between the test and reference products and its 90% CI. Geometric Coefficient of variation was provided as percentage.
Time Frame: 0.75, 0.5, 0.25 hours predose and 0.08, 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 2, 3, 4, 6, 8 10, 14, 16, 20 and 24 hours postdose in each treatment period
Population: Pharmacokinetic analysis set1 (PKAS1) included all randomized participants who completed both periods, had no major protocol deviations concerning pharmacokinetics, excluding those with baseline nicotine concentration greater than (>) 5 percent (%) of individual highest observed plasma nicotine concentration (Cmax) for either period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter(ng*hr/mL)
Groups:
- Prototype Mini Lozenges: Participants randomized to receive a single dose of Treatment A: 2 mg of Prototype Mini Lozenge administered orally in either Treatment Period 1 (on Day 1) or Treatment Period 2 (Day 5 to 7). All these doses were administered after an overnight fast of at least 10 hours in each period. Participants were confined in the study facility for approximately 60 hours during each treatment period (for 36 hours predose and for 24 hours postdose) with abstinence from smoking during which they were subjected to random measurements of expired CO to confirm abstinence (CO levels must have been <= 10 ppm throughout the treatment period).
- Nicorette Mini Lozenges: Participants randomized to receive a single dose of Treatment B: 2 mg of Nicorette Mini lozenge administered orally in either Treatment Period 1 (on Day 5 to 7) or Treatment Period 2 (Day 1). All these doses were administered after an overnight fast of at least 10 hours in each period. Participants were confined in the study facility for approximately 60 hours during each treatment period (for 36 hours predose and for 24 hours postdose) with abstinence from smoking during which they were subjected to random measurements of expired CO to confirm abstinence (CO levels must have been <= 10 ppm throughout the treatment period).
Arm/Group | Prototype Mini Lozenges | Nicorette Mini Lozenges
Number analyzed (Participants) | 25 | 25
nanograms*hours per milliliter(ng*hr/mL) | 15.39 (39.40) | 16.19 (40.10)
Statistical Analysis 1: Comparison: Prototype Mini Lozenges vs Nicorette Mini Lozenges; Test type: Equivalence — Bioequivalence was determined if the 90% CIs of the GMRs for AUC0-t fell completely within the 0.80 - 1.25 range; Geometric mean ratio = 0.95, 90% CI 2-sided [0.91 to 1.00] — GMR= (Prototype mini Lozenge/ Nicorette mini Lozenge)

2. Primary Outcome: Assessment of Bioequivalence of Prototype Mini Lozenges With Nicorette Mini Lozenge by Measuring Area Under the Plasma Concentration Versus Time Curve Calculated From Time Zero to Infinity (AUC [(0-inf])
Description: Bioequivalence of prototype mini lozenges with nicorette mini lozenge was assessed by measuring AUC(0-inf). AUC(0-inf) = AUC0-t + (Clast/kel), where, AUC0-t= area under the plasma concentration versus time curve from time zero to time t; Clast= last observed/measured plasma concentration and kel= elimination rate constant. A linear mixed-effects model was fit to the natural log (ln)-transformed PK variable (AUC[0-inf]), as the dependent variable, and treatment, period, and sequence as fixed effects. Participant nested within sequence was a random effect. The treatment difference and its 90% CI were exponentiated to obtain the GMR between the test and reference products and its 90% CI. Geometric Coefficient of variation was provided as percentage.
Time Frame: as for outcome 1
Population: Analysis performed on PKAS1, that included all randomized participants who completed both periods, had no major protocol deviations concerning pharmacokinetics, excluding those with baseline nicotine concentration > 5% of individual Cmax for either period. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Prototype Mini Lozenges | Nicorette Mini Lozenges
Number analyzed (Participants) | 25 | 25
ng*hr/mL | 16.53 (39.50) | 17.38 (40.20)
Statistical Analysis 1: Comparison: Prototype Mini Lozenges vs Nicorette Mini Lozenges; Test type: Equivalence — Bioequivalence was determined if the 90% CIs of the GMRs for AUC(0-inf) fell completely within the 0.80 - 1.25 range; Geometric Mean Ratio = 0.94, 90% CI 2-sided [0.89 to 1.00] — GMR = (Prototype mini Lozenge/Nicorette mini Lozenge)

3. Primary Outcome: Assessment of Bioequivalence of Prototype Mini Lozenges With Nicorette Mini Lozenge by Measuring Maximum Observed Plasma Nicotine Concentration (Cmax)
Description: Blood samples were collected at designated timepoints. Bioequivalence of prototype mini lozenges with nicorette mini lozenge was assessed by measuring Cmax that was taken directly from bioanalytical data. Geometric Coefficient of variation was provided as percentage. A linear mixed-effects model was fit to the natural log (ln)-transformed PK variable (Cmax) as the dependent variable, and treatment, period, and sequence as fixed effects. Participant nested within sequence was a random effect. The treatment difference and its 90% CI were exponentiated to obtain the GMR between the test and reference products and its 90% CI. Geometric Coefficient of variation was provided as percentage.
Time Frame: as for outcome 1
Population: Analysis performed on PKAS1, that included all randomized participants who completed both periods, had no major protocol deviations concerning pharmacokinetics, excluding those with baseline nicotine concentration > 5% of individual Cmax for either period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Prototype Mini Lozenges | Nicorette Mini Lozenges
Number analyzed (Participants) | 25 | 25
nanograms per milliliter | 4.41 (32.10) | 4.89 (33.80)
Statistical Analysis 1: Comparison: Prototype Mini Lozenges vs Nicorette Mini Lozenges; Test type: Equivalence — Bioequivalence was determined if the 90% CIs of the GMRs for Cmax fell completely within the 0.80 - 1.25 range; Geometric Mean Ratio = 0.89, 90% CI 2-sided [0.82 to 0.98] — GMR = (Prototype mini Lozenge/Nicorette mini Lozenge)

4. Secondary Outcome: Comparison of Prototype Mini Lozenges With Nicorette Mini Lozenge by Measuring Time of Maximum Plasma Nicotine Concentration (Tmax)
Description: Tmax was defined as the time to maximum plasma nicotine concentration. If the maximum value occurred at more than one time point, Tmax was defined as the first time point with this value.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Prototype Mini Lozenges | Nicorette Mini Lozenges
Number analyzed (Participants) | 25 | 25
hour | 1.02 [0.83 to 1.28] | 1.02 [0.85 to 1.26]

5. Secondary Outcome: Comparison of Prototype Mini Lozenges With Nicorette Mini Lozenge by Measuring Apparent Elimination Half-Life (t1/2)
Description: t1/2 was defined as apparent elimination half-life that was calculated as t1/2 = ln(2) / Kel, where Kel= elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Full Range); unit: hour
Arm/Group | Prototype Mini Lozenges | Nicorette Mini Lozenges
Number analyzed (Participants) | 25 | 25
hour | 3.64 [1.53 to 14.39] | 3.46 [1.46 to 14.84]

6. Secondary Outcome: Comparison of Prototype Mini Lozenges With Nicorette Mini Lozenge by Measuring Apparent Elimination Rate Constant for Plasma Nicotine (Kel)
Description: kel was defined as apparent elimination rate constant for plasma nicotine that was calculated as negative of the slope of a linear regression of the log(concentration)- time for all concentrations > lower limit of quantification.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Full Range); unit: fraction per hour
Arm/Group | Prototype Mini Lozenges | Nicorette Mini Lozenges
Number analyzed (Participants) | 25 | 25
fraction per hour | 0.28 [0.05 to 0.45] | 0.28 [0.05 to 0.48]

7. Secondary Outcome: Number of Participants With Clinically Significant Change in Laboratory Test Values
Description: Haematological, biochemistry and urinalysis parameters were analyzed. Clinical significance was judged by the investigator based upon the out of range values of standard range set for each parameter.
Time Frame: From signing of the informed consent form until 5 days after last administration of study drug (up to Day 13)
Population: Safety population was defined as all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Prototype Mini Lozenges | Nicorette Mini Lozenges | All Treatment Combined
Number analyzed (Participants) | 46 | 44 | 46
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form until 5 days after last administration of study drug (up to Day 13)
Description: Safety population: all randomized participants who received at least one dose of study medication. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported. A participant with multiple occurrences of AEs counted once in AE category. A participant with multiple AEs within a primary system organ class was counted once in system organ class.
Arm/Group | Prototype Mini Lozenges | Nicorette Mini Lozenges | All Treatment Combined
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 13/46 | 15/44 | 23/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prototype Mini Lozenges (N=46) | Nicorette Mini Lozenges (N=44) | All Treatment Combined (N=46)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Oral discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tongue discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 2 (2) | 2 (3)
Vessel puncture site pain (General disorders) | 3 (3) | 4 (4) | 7 (7)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3) | 5 (8)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT03541044/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT03541044/SAP_001.pdf